CLINICAL TRIAL: NCT02899897
Title: Place of Echocardiography in IV Fluid Therapy in Patients With Septic Shock and Left Ventricular Systolic Dysfunction: a Multicentre Prospective Study
Brief Title: Place of Echocardiography in IV Fluid Therapy in Patients With Septic Shock and Left Ventricular Systolic Dysfunction
Acronym: DYSPRED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-37 Dr Zogheib
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Shock, Septic; Ventricular Dysfunction, Left
Keywords: echocardiography
MeSH Terms: conditions — Shock, Septic; Ventricular Dysfunction, Left | interventions — Echocardiography; Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: echocardiography in IV fluid therapy

SUMMARY:
IV fluid therapy remains an essential haemodynamic objective in the treatment strategy of septic shock. Left ventricular systolic dysfunction secondary to sepsis is observed in 40% and up to 65% of the population concerned. However, the capacity of the various indices to predict the response to IV fluid therapy in septic shock with left ventricular systolic dysfunction have not been clearly defined. Measurement of parameters reflecting filling pressures during transthoracic echocardiography (TTE) is one of the methods used to evaluate cardiac function and estimate the filling reserve, but with no strong evidence. Right heart catheterization with determination of cardiac output by pulmonary thermodilution can also be used to measure the various parameters commonly used to predict the response to IV fluid therapy. Very few data are available with no reliable and clinically relevant data in this population with septic shock and left ventricular systolic dysfunction (LVEF ≤ 40%) and the response to IV fluid therapy monitored by dynamic indices obtained by transpulmonary thermodilution and right heart catheterization. Consequently, the capacity of the various indices of preload dependence to predict the response to IV fluid therapy in septic shock with left ventricular systolic dysfunction remains difficult to define.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock with cardiovascular dysfunction despite norepinephrine,
* Left ventricular systolic dysfunction defined by transthoracic echocardiography and LVEF ≤ 40%
* Fluid challenge decided by the patient's attending physician according to the optimization of cardiac output in septic shock protocol,
* IV fluid therapy with 500 ml of crystalloid solution.
* Haemodynamic monitoring decided by the patient's referring physician not involved in the study, according to the department's usual practice by transthoracic echocardiography and thermodilution monitoring.
* Sedated, on mechanical ventilation, and adapted to the ventilator.
* Patients who have received oral information and written documentation (with a copy filed in the medical records) on awakening.
* The trusted person designated for each patient has received the same oral and written information.

Exclusion Criteria:

Patients under the age of 18 years, pregnant women, patients under judicial protection or deprived of their freedom, Amputation of one or both lower limbs Contraindication to passive leg raising (e.g.: severe IC, etc.), Cardiac tamponade or aortic dissection with uncontrolled active bleeding. No indication for IV fluid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Response to IV fluid therapy | 90 minutes
  defined by an increase in stroke volume by more than 15% of its baseline value measured by thermodilution.

CONTACTS AND LOCATIONS:
Overall Officials: Elie ZOGHEIB, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France